CLINICAL TRIAL: NCT00045773
Title: Treatment Outcome of Vascular Depression
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Duke University (Other)
Responsible Party: Principal Investigator, Yvette Sheline, Penn Faculty - McLure Professor, University of Pennsylvania
Other Study IDs: R01MH060697 (NIH); R01MH060697 (NIH); DATR A4-GPX
Record Dates: First submitted 2002-09-09; First posted 2002-09-11 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Sertraline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — 50 - 200mg, once per day for 12 weeks.
  Other Names: Zoloft

SUMMARY:
This 12-week study will evaluate the effectiveness of sertraline (Zoloft®) for treatment of depression associated with small vascular lesions in the brain (vascular depression).

DETAILED DESCRIPTION:
Major late life depression (LLD) is an important health problem with a large and growing number of affected individuals. A significant subset of patients with LLD, particularly those with vascular depression, have abnormalities in certain parts of the brain that are evident on MRI scans and may be associated with poor acute and long-term response to antidepressant treatment. Studies have also indicated that LLD patients frequently have frontal lobe dysfunction. A longitudinal study with the antidepressant nortriptyline has demonstrated that frontal lobe dysfunction is associated with poor acute response and a greater risk for recurrence of LLD. However, it is not known if this finding applies to other antidepressants. This study will be the first clinical trial to simultaneously test the effects of specific brain and psychological factors on course of response, remission rate, and other measures of health outcomes in people with LLD.

Participants are treated with sertraline for 12 weeks. During this period, participants undergo cognitive testing, MRI, electrocardiogram (EKG), and laboratory tests. Study visits occur every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 60+
2. DSM-IV criteria for MDD
3. Hamilton Depression Rating Scale score >18
4. No MRI contraindications, e.g. foreign metallic implants, pacemaker
5. Medication free of any psychotropic drug except as otherwise noted for set washout period (see D.2.1)
6. Mini Mental Status Exam score <21
7. No unstable medical disorders (requiring immediate medical attention)
8. Ability to give informed consent
9. English speaking

Exclusion Criteria:

1. Age <60
2. Does not meet DSM-IV criteria for MDD
3. Hamilton Depression Rating Scale score <18
4. MRI contraindications e.g. foreign metallic implants, pacemaker
5. Psychotropic drug use other than zolpidem and lorazepam, prn within 2 weeks of entry
6. Mini Mental Status Exam score >21, or known primary neurological disorders including Dementia of the Alzheimer type, Parkinson's Disease, multiple sclerosis, seizure disorder.
7. Unstable medical disorders, uncorrected hypothyroidism, or any condition that in the investigators opinion makes the patients unsuitable for a trial
8. Cannot give informed consent
9. Does not speak English

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 60+ with major depression.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2001-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette I. Sheline, M.D., Principal Investigator — Washington University Psychiatrist; Murali Doraiswamy, M.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Sheline YI, Black KJ, Lin DY, Christensen GE, Gado MH, Brunsden BS, Vannier MW. Stereological MRI volumetry of the frontal lobe. Psychiatry Res. 1996 Oct 7;67(3):203-14. doi: 10.1016/0925-4927(96)02831-4. PMID 8912959
- [Background] Sheline Y, Loenze E, Cross D, et al., (1996) Quantifying white matter lesions in elderly women with depression. Presented at the Annual Meeting of the American College of Neuropsychopharmacology, San Juan, Puerto Rico.
- [Background] Sheline YI, Freedland KE, Carney RM. How safe are serotonin reuptake inhibitors for depression in patients with coronary heart disease? Am J Med. 1997 Jan;102(1):54-9. doi: 10.1016/s0002-9343(96)00374-9. PMID 9209201
- [Background] Sheline Y.I. Neuroanatomical changes associated with unipolar major depression. The Neuroscientist 4:331-334, 1998
- [Result] Sheline YI, Price JL, Vaishnavi SN, Mintun MA, Barch DM, Epstein AA, Wilkins CH, Snyder AZ, Couture L, Schechtman K, McKinstry RC. Regional white matter hyperintensity burden in automated segmentation distinguishes late-life depressed subjects from comparison subjects matched for vascular risk factors. Am J Psychiatry. 2008 Apr;165(4):524-32. doi: 10.1176/appi.ajp.2007.07010175. Epub 2008 Feb 15. PMID 18281408
- [Result] Sheline YI, Barch DM, Garcia K, Gersing K, Pieper C, Welsh-Bohmer K, Steffens DC, Doraiswamy PM. Cognitive function in late life depression: relationships to depression severity, cerebrovascular risk factors and processing speed. Biol Psychiatry. 2006 Jul 1;60(1):58-65. doi: 10.1016/j.biopsych.2005.09.019. Epub 2006 Jan 18. PMID 16414031
- [Derived] Sheline YI, Pieper CF, Barch DM, Welsh-Bohmer K, McKinstry RC, MacFall JR, D'Angelo G, Garcia KS, Gersing K, Wilkins C, Taylor W, Steffens DC, Krishnan RR, Doraiswamy PM. Support for the vascular depression hypothesis in late-life depression: results of a 2-site, prospective, antidepressant treatment trial. Arch Gen Psychiatry. 2010 Mar;67(3):277-85. doi: 10.1001/archgenpsychiatry.2009.204. PMID 20194828
- See also: Volunteer for Health with Washington University School of Medicine — https://vfh.wustl.edu/
- See also: Washington University School of Medicine Psychiatry Department — http://www.psychiatry.wustl.edu